CLINICAL TRIAL: NCT04681053
Title: Efficacy and Safety of Inhaled Ivermectin in the Treatment of SARS-COV-2 (COVID-19)
Brief Title: Inhaled Ivermectin and COVID-19
Acronym: CCOVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Elbendary, Professor of Tropical Medicine and Hepatogastroenterology, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R.20.11.1090.R1
Record Dates: First submitted 2020-12-16; First posted 2020-12-23 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
Keywords: COVID; Ivermectin; Inhalation; Antiviral; safety
MeSH Terms: conditions — COVID-19; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: All current study participants will be classified into 4 equal groups
  : Group (A) received both oral and inhaled ivermectin in addition to the standard of care.
  Group (B)received inhaled ivermectin only Group (C) received oral ivermectin in addition to the standard of care, Group (D) received the current standard of care only
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group (A) received both oral and inhaled ivermectin in addition to the standard of care. (Active Comparator): use oral and inhaled ivermectin
  Interventions: Drug: Ivermectin Powder
- B) received oral ivermectin in addition to the standard of care (Active Comparator): receive oral ivermectin
  Interventions: Drug: Ivermectin Powder
- c) received inhaled ivermectin in addition to the standard of care (Active Comparator): received inhaled ivermectin
  Interventions: Drug: Ivermectin Powder
- Group (d) received the current standard of care only (No Intervention): received standard of care only

INTERVENTIONS:
Drug: Ivermectin Powder — - Administration through inhalation (6mg) BID for 3 days
  Other Names: Direct antiviarl agents
  Arms: B) received oral ivermectin in addition to the standard of care; Group (A) received both oral and inhaled ivermectin in addition to the standard of care.; c) received inhaled ivermectin in addition to the standard of care

SUMMARY:
Coronavirus disease-19 is global healthcare crisis. Till May 20, 2020, there were approximately 4,789,205 cases and 318,789 related mortalities were identified globally. This dramatic situation led to healthcare service collapse in many countries. Each country developed its own action plan depending on healthcare expertise and the available resources. There is no definitive therapy for Coronavirus disease-19 up till now. Many current and investigational drugs are used nowadays. Recent reports suggest a beneficial role of Ivermectin in the management of Coronavirus disease-19. A notice that necessitates further clinical studies.

The aim of this study is to assess the efficacy and safety of the usage of inhaled ivermectin in the management of Coronavirus disease-19.

DETAILED DESCRIPTION:
Coronavirus disease-19 (COVID-19) is a pandemic disease which is caused by the SARS-CoV2 virus. It is one of the biggest single-stranded RNA viruses. SARS-CoV2 Viral polyproteins are responsible for viral replication and transcription while its protease enzymes are responsible for polypeptides cleaving and immune system blockage. They are considered to be an important therapeutic target.

Host immunological response against SARS-CoV2 could affect the disease outcome. Patients requiring ICU admission have higher levels of interleukins 6 - 10, tumor necrosis factor α (TNF-α), and fewer CD4+ and CD8+ T cells. The level of cytokines and lymphopenia is associated with pulmonary damage and respiratory distress.

Till now, there is no definitive therapy for COVID-19. Multiple current and investigational drugs are used such as Hydroxychloroquine, lopinavir/ritonavir, and Remdesivir.

Ivermectin: A potent anti-parasitic drug has shown to have an in-vitro antiviral activity against a broad range of viruses. It inhibits the interaction between the human immunodeficiency virus-1 (HIV-1) integrase protein (IN) and the importin (IMP) α/β1. But on the other hand, Ivermectin showed limited efficacy against DENV in phase III clinical trial that was done in Thailand in 2014-2017. Recent Studies proved the In-vitro effect and "subsequently" the possible therapeutic role of Ivermectin in the management of SARS-CoV2.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age above 18
* Test positive for COVID-19 using Reverse transcription polymerase chain reaction (RT-PCR) prior to the start of study.
* Willing to participate in the study
* Mild to moderate severity index according to the WHO criteria

Exclusion Criteria:

* Hypersensitivity to the study drug.
* History of co-morbid conditions such as: uncontrolled hypertension and diabetes, retinal problems and chronic liver and renal disease.
* Women who are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-02-25 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of virological cure by Rt -PCR for COVID -19 using ivermectin when compared to standard treatment | througout the study completion up to one year(for every case must be done after 2 weeks from the start of treatment).
  All PCR for COVID-19 must be negative

SECONDARY OUTCOMES:
resolution of pneumonia | througout the study completion up to one year (for every case must be done after 2 weeks from the start of treatment).
  The score severity index of pneumonia will be measured before and after receiving treatment by computed tomography (CT)(index from 0-20)increasing the index means increase severity.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud El-Bendary, M.D, Principal Investigator — Mansoura University- Faculty of Medicine
Locations (1):
- Mansoura Faculty of Medicine, Al Mansurah, Dakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: No